CLINICAL TRIAL: NCT07173010
Title: Pediatric Arthropathy Beyond Inflammation: Clinical Spectrum and Diagnostic Approach at Assiut University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nora Ammar Shawket, Principal investigator, Assiut University
Other Study IDs: Non inflammatory arthropathy
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mucopolysaccharidoses; Progressive Pseudorheumatoid Dysplasia; Farber Disease; Osteogenesis Imperfecta; Infantile Systemic Hyalinosis; Idiopathic Multicentric Osteolysis
MeSH Terms: conditions — Mucopolysaccharidoses; Arthropathy, progressive pseudorheumatoid, of childhood; Farber Lipogranulomatosis; Osteogenesis Imperfecta; Hyaline Fibromatosis Syndrome; Osteolysis, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the most common underlying causes of non-inflammatory arthropathy in children presenting to Assiut University Children Hospital for through clinical evaluation, laboratory testing, and imaging, in order to improve diagnostic precision, guide appropriate management, and distinguish these conditions from inflammatory joint diseases.

DETAILED DESCRIPTION:
Arthropathy refers to any disease or abnormal condition of a joint. It includes both inflammatory ( arthritis) and non-inflammatory types. Arthritis involves joint inflammation with symptoms such as pain, swelling, and stiffness, along with elevated inflammatory markers. In contrast, non-inflammatory arthropathy may mimic arthritis but lacks signs of inflammation and typically shows normal inflammatory markers.

Non inflammatory arthropathy can closely mimic juvenile idiopathic arthritis (JIA), leading to frequent misdiagnosis and inappropriate treatment.

These disorders are sometimes incorrectly diagnosed and treated as JIA, patients often do not respond to immunosuppressive treatment, leading to poor compliance, disease progression, and unnecessary exposure to potentially harmful medications.

A high index of suspicion, detailed clinical evaluation, and appropriate imaging are essential to distinguish these mimics from true inflammatory arthritis.

Here's a breakdown of some conditions categorized as non-inflammatory arthropathies:

Mucopolysaccharidoses (MPS) are rare inherited metabolic disorders caused by enzyme deficiencies that impair the breakdown of glycosaminoglycans (GAGs), leading to their accumulation and progressive tissue and organ damage. Patients often present with arthropathy ,joint stiffness alongside hallmark features such as skeletal abnormalities, developmental delays, intellectual disability, cardiac issues, corneal clouding, hearing loss, short stature, dysostosis multiplex, and coarse facial features.However Some attenuated forms of mucopolysaccharidoses (MPS), particularly MPS I (Scheie syndrome), MPS II (attenuated Hunter syndrome), and MPS VI (Maroteaux-Lamy syndrome), may present predominantly with joint stiffness and contractures without significant systemic or cognitive involvement.

Progressive Pseudorheumatoid Dysplasia (PPRD) is a rare autosomal recessive skeletal disorder caused by mutations in the WISP3 gene, crucial for joint cartilage development and function. It leads to progressive degeneration of articular cartilage, primarily affecting the interphalangeal joints. Patients typically present with painless, progressive joint stiffness and enlargement without inflammation, joint contractures, gait abnormalities, and spinal deformities such as scoliosis or kyphosis, resulting in abnormal posture and muscle weakness-related morbidities.

Camptodactyly-Arthropathy-Coxa Vara-Pericarditis (CACP) syndrome is a rare autosomal recessive disorder characterized by congenital or early-onset camptodactyly, non-inflammatory arthropathy with synovial hyperplasia, progressive coxa vara deformity of the hip, and non-inflammatory pericarditis. Joint effusions are typically cool and unresponsive to anti-inflammatory treatments.

Idiopathic Multicentric Osteolysis is a rare autosomal dominant skeletal disorder characterized by progressive osteolysis primarily affecting the carpal and tarsal bones, leading to joint deformities, pain, and mobility loss. Typically presenting in childhood, patients experience arthritic-like episodes, progressive deformities, osteolytic changes on imaging, and varying degrees of disability. Associated features may include short stature, muscle weakness, cardiovascular abnormalities, chronic renal failure, as well as occasional mental retardation and minor facial anomalies.

Infantile Systemic Hyalinosis (ISH) is a rare autosomal recessive fibromatosis caused by mutations in the ANTXR2 (CMG2) gene, resulting in widespread hyaline material deposition in multiple tissues including skin, joints, and internal organs. Clinically, ISH presents with painful joint contractures which may lead to arthrogryposis-like appearance (multiple joint contractures), Progressive stiffness and fixed flexion deformities develop especially in knees, elbows, hips, and fingers ,Limited range of motion,subcutaneous nodules, gingival hypertrophy, osteopenia, failure to thrive, protein-losing enteropathy with diarrhea, and recurrent infections.

Farber disease is a rare, fatal autosomal recessive metabolic disorder caused by mutations in the ASAH1 gene, leading to deficient acid ceramidase enzyme activity and subsequent ceramide accumulation in tissues. Affected children typically present with progressive painful joint stiffness, limited motion, contractures, subcutaneous nodules, and hoarseness due to laryngeal involvement, which can result in breathing difficulties.

Osteogenesis imperfecta (OI) is a genetic connective tissue disorder caused by mutations in the COL1A1 and COL1A2 genes, leading to defective type I collagen synthesis. Characterized by brittle bones with increased fracture risk and low bone density,Skeletal deformities and recurrent fractures contribute to abnormal joint mechanics, resulting in arthropathy, stiffness, reduced mobility, and functional impairment over time. OI also presents with blue sclerae, dentinogenesis imperfecta, short stature, and adult-onset hearing loss. Cardiovascular manifestations such as valvular insufficiencies and aortic root dilation have been reported. Milder symptoms include joint laxity, easy bruising, hernias, and hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children up to 18 years at diagnosis.
* Patients presents with picture of non inflammatory arthropathy as joint deformity, stiffness and skeletal abnormality (arthropathy) with normal inflammatory markers

Exclusion Criteria:

* Patients more than 18years.
* Patients presents with painful,hot, tender or red joints (Arthritis) associated with elevated inflammatory markers .

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will include all pediatric patients presented with non inflammatory arthropathy based on clinical manifestations, laboratory investigations and imaging up to age of 18 years in the last 3 years (retrospective) and those who will present newly through a duration of one year (preospective). They will be recruited from the inpatient and outpatient clinic of Allergy, Immunology and Rheumatology department at Assuit University Children's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To diagnose most common causes of non inflammatory arthropathy | 1year
  To identify the most common underlying causes of non-inflammatory arthropathy in children presenting to Assiut University Children Hospital for through clinical evaluation, laboratory testing, and imaging, in order to improve diagnostic precision, guide appropriate management, and distinguish these conditions from inflammatory joint diseases

SECONDARY OUTCOMES:
To avoid misdiagnosis as inflammatory arthropathy | 1year
  To Avoid use of unnecessary treatment in patients with non inflammatory arthropathy who wrongly diagnosed as inflammatory arthropathy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Porell FW, Miltiades HB. Disability outcomes of older Medicare HMO enrollees and fee-for-service Medicare beneficiaries. J Am Geriatr Soc. 2001 May;49(5):615-31. doi: 10.1046/j.1532-5415.2001.49123.x. PMID 11380756
- [Background] Emerson GG, Segal SS. Endothelial cell pathway for conduction of hyperpolarization and vasodilation along hamster feed artery. Circ Res. 2000 Jan 7-21;86(1):94-100. doi: 10.1161/01.res.86.1.94. PMID 10625310
- [Background] Sands MS. Farber disease: understanding a fatal childhood disorder and dissecting ceramide biology. EMBO Mol Med. 2013 Jun;5(6):799-801. doi: 10.1002/emmm.201302781. Epub 2013 May 13. No abstract available. PMID 23666771
- [Background] Maatallah K, Boussaa H, Lassoued Ferjani H, Kaffel D, Hamdi W. Progressive pseudorheumatoid dysplasia: A rare entity mimicking juvenile idiopathic arthritis. Clin Case Rep. 2021 Aug 16;9(8):e04670. doi: 10.1002/ccr3.4670. eCollection 2021 Aug. PMID 34430024
- [Background] Muenzer J. Overview of the mucopolysaccharidoses. Rheumatology (Oxford). 2011 Dec;50 Suppl 5:v4-12. doi: 10.1093/rheumatology/ker394. PMID 22210669
- [Background] Khan SA, Peracha H, Ballhausen D, Wiesbauer A, Rohrbach M, Gautschi M, Mason RW, Giugliani R, Suzuki Y, Orii KE, Orii T, Tomatsu S. Epidemiology of mucopolysaccharidoses. Mol Genet Metab. 2017 Jul;121(3):227-240. doi: 10.1016/j.ymgme.2017.05.016. Epub 2017 May 26. PMID 28595941
- [Background] Ablin DS. Osteogenesis imperfecta: a review. Can Assoc Radiol J. 1998 Apr;49(2):110-23. PMID 9561014
- [Background] Carnevale A, Canun S, Mendoza L, del Castillo V. Idiopathic multicentric osteolysis with facial anomalies and nephropathy. Am J Med Genet. 1987 Apr;26(4):877-86. doi: 10.1002/ajmg.1320260415. PMID 3591830
- [Background] Tasar M, Eyileten Z, Kasimzade F, Ucar T, Kendirli T, Uysalel A. Camptodactyly-arthropathy-coxa vara-pericarditis (CACP) syndrome. Turk J Pediatr. 2014 Nov-Dec;56(6):684-6. PMID 26388606
- [Background] Bhavani GS, Shah H, Shukla A, Dalal A, Girisha KM. Progressive Pseudorheumatoid Dysplasia. 2015 Nov 25 [updated 2020 Dec 23]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK327267/ PMID 26610319
- [Background] Al-Mayouf SM. Noninflammatory disorders mimic juvenile idiopathic arthritis. Int J Pediatr Adolesc Med. 2018 Mar;5(1):1-4. doi: 10.1016/j.ijpam.2018.01.004. Epub 2018 Feb 24. PMID 30805524
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases. Arthritis . Bethesda (MD): National Institutes of Health; 2022 Nov. — https://www.niams.nih.gov/health-topics/arthritis